CLINICAL TRIAL: NCT01151540
Title: A Long Term Extension Study of E2080 in Lennox-Gastaut Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2080-J081-305
Record Dates: First submitted 2010-06-14; First posted 2010-06-28 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-03

CONDITIONS: Lennox-Gastaut Syndrome
Keywords: Epilepsy; Seizures
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epilepsy; Seizures | interventions — rufinamide

ARMS (1):
- Rufinamide (Experimental): Ralfinamide was administered orally twice daily after breakfast and dinner. Participants on placebo in Study 304 were titrated over to rufinamide within 2 weeks during the Conversion Period. As a general rule, the dose of rufinamide at the end of the Conversion Period was maintained throughout the Maintenance Period.
  Interventions: Drug: Rufinamide

INTERVENTIONS:
Drug: Rufinamide — The target dosage is approximately 45 mg/kg/day, taken orally twice a day.
  Other Names: E2080, BANZEL

SUMMARY:
To investigate the safety of long term administration of E2080 in the patients with Lennox-Gastaut syndrome who completed the E2080-J081-304 Study.

ELIGIBILITY:
Inclusion criteria:

1. Participants who have completed the evaluation of Week 12 of the E2080-J081-304 study.
2. Male participants with reproductive ability and female participants with child-bearing potential, or their partners, had to be able to take medically appropriate contraceptive measures.
3. Participants who have provided a written informed consent to participate in this clinical trial until the evaluation of week 12 of the E2080-J081-304 study.
4. Participants who had a family member or a caregiver capable of recording the reporting diary, providing participant information necessary for the study, assisting treatment compliance, and accompanying the participant on scheduled visit days during the study period.

Exclusion criteria:

1. Participants who were judged by the investigator that they are unfit to participate in this clinical study for safety reasons based on the information up to the evaluation of week 12 of the E2080-J081-304 Study.
2. Participants who were judged by the investigator that they are likely to become non-compliant with administration during the clinical trial period.
3. Participants who were judged by the investigator that they were unfit to participate in this clinical trial.

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Takano, Study Director — Neuroscience Clinical Development Section. JAC PCU. Eisai Co., Ltd.
Locations (23):
- Japan (23):
  - Nagoya, Aichi-ken
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Yokohama, Kanagawa
  - Goshi^shi, Kumamoto
  - Iwanuma-shi, Miyagi
  - Ōmura, Nagasaki
  - Nara, Nara
  - Niigata, Niigata
  - Yufu-shi, Oita Prefecture
  - Neyagawa, Osaka
  - Osaka, Osaka
  - Suita-shi, Osaka
  - Moriyama-shi, Shiga
  - Shizuoka, Shizuoka
  - Kodaira, Tokyo
  - Kokubunji-shi, Tokyo
  - Shinjuku, Tokyo
  - Toyoma-shi, Toyama
  - Okayama

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who successfully completed Study 304 were enrolled into this study.
Period: Overall Study
Arm/Group | Rufinamide
Started | 54
Completed | 41
Not Completed | 13
Not completed — Other | 2
Not completed — Adverse event, non-fatal | 4
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all treated participants.
Arm/Group | Rufinamide
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15 (6.8)
Age, Customized [Number; unit: Participants]
  ≥4 to <12 years | 22
  ≥12 to <17 years | 11
  ≥17 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability of Rufinamide
Description: Safety was assessed by monitoring and recording all adverse events (AEs), serious adverse events (SAEs), clinical laboratory tests, blood pressure, pulse rate, physical examination, and 12-lead electrocardiogram (ECG). Treatment-emergent adverse events (TEAEs) were defined as AEs that started on or after the date and time of administration of first dose of test drug, but not later than 30 days after discontinuation from the study, or if the AE was present prior to the administration of the first dose of test drug and increased in National Cancer Institute Common Toxicity Criteria (NCI CTC version 3.0) grade during the study or 30 days after discontinuation from the study. AEs were considered serious if it resulted in; death, was life-threatening, hospitalization/prolonged hospitalization, persistent or significant disability/incapacity, or a congenital anomaly/birth defect.
Time Frame: From date of first dose up to 30 days after the last dose of study treatment, up to approximately 2 years 10 months
Population: Safety analysis set included all treated participants.
Measure: Number; unit: Participants
Arm/Group | Rufinamide
Number analyzed (Participants) | 54
Participants
  TEAEs | 54
  Treatment-related TEAEs | 38
  SAEs | 9
  Treatment-related SAEs | 2
  AEs leading to study drug withdrawal | 3
  AEs leading to study drug dose reduction | 12

2. Secondary Outcome: Percent Change in Tonic-Atonic Seizure Frequency From Baseline (Per 28 Days)
Description: The sum of the frequencies of tonic seizures and atonic seizures was defined as the "tonic-atonic seizure frequency". The percent change in tonic-atonic seizure frequency was calculated using the tonic-atonic seizure frequency per 28 days of the Observation Period in Study 304 as the baseline and the tonic-atonic seizure frequency at Weeks 12, 24, 32, 40, 52 and Week 52 Last Observation Carried Forward (LOCF) as the post-treatment value. Percentage change in tonic - atonic seizure frequency was calculated as follows: [100 x (post-treatment value - baseline)/ baseline]. The frequency of epileptic seizures was recorded in the seizure diary by the recorder. Seizure frequency was counted based on the classification established by the International League Against Epilepsy (ILAE). The diary recorder monitored the participant and recorded the seizure diary in a consistent manner, and continued these practices throughout the study period.
Time Frame: Baseline (Observation period in Study 304), Week 12, Week 24, Week 32, Week 40, Week 52 and Week 52 LOCF
Population: Efficacy Analysis Set included all participants with evaluable efficacy data.
Measure: Median (Full Range); unit: Percent Change in Seizure Frequency
Arm/Group | Rufinamide
Number analyzed (Participants) | 46
Percent Change in Seizure Frequency
  Percent Change in Week 12 | -39.3 [-100 to 125.2]
  Percent Change in Week 24: number analyzed (Participants) | 43
  Percent Change in Week 24 | -40.6 [-100 to 85.7]
  Percent Change in Week 32: number analyzed (Participants) | 42
  Percent Change in Week 32 | -46.8 [-100 to 75]
  Percent Change in Week 40: number analyzed (Participants) | 41
  Percent Change in Week 40 | -47.6 [-100 to 833.2]
  Percent Change in Week 52: number analyzed (Participants) | 40
  Percent Change in Week 52 | -36.05 [-100 to 101.7]
  Percent Change in Week 52 LOCF | -39.25 [-100 to 101.7]

3. Secondary Outcome: Percent Change in the Total Seizure Frequency From Baseline (Per 28 Days)
Description: Percent change in the total seizure frequency (per 28 days) was calculated using the total seizure frequency per 28 days of the Observation Period of Study 304 as the baseline and the total seizure frequency per 28 days at Weeks 12, 24, 32, 40, 52 and Week 52 LOCF as the post-treatment value. Percentage change in total seizure frequency was calculated as follows: [100 x (post-treatment value - baseline)/ baseline].
Time Frame: Baseline (Observation period in Study 304), Week 12, Week 24, Week 32, Week 40, Week 52 and Week 52 LOCF
Population: Efficacy Analysis Set included all participants with evaluable efficacy data.
Measure: Median (Full Range); unit: Percent Change in Seizure Frequency
Arm/Group | Rufinamide
Number analyzed (Participants) | 46
Percent Change in Seizure Frequency
  Percent Change in Week 12: number analyzed (Participants) | 45
  Percent Change in Week 12 | -47.7 [-100 to 101.5]
  Percent Change in Week 24: number analyzed (Participants) | 43
  Percent Change in Week 24 | -48.9 [-97 to 116.6]
  Percent Change in Week 32: number analyzed (Participants) | 42
  Percent Change in Week 32 | -50.6 [-90.8 to 209.2]
  Percent Change in Week 40: number analyzed (Participants) | 41
  Percent Change in Week 40 | -52 [-95.5 to 833.2]
  Percent Change in Week 52: number analyzed (Participants) | 40
  Percent Change in Week 52 | -47.35 [-94.3 to 340.8]
  Percent Change in Week 52 LOCF | -46.3 [-100 to 340.8]

4. Secondary Outcome: Percent Change in the Frequency of Seizures Other Than Tonic-Atonic Seizures
Description: Percent change in the frequency of seizures other than tonic-atonic seizures (per 28 days) was calculated using the total seizure frequency per 28 days of the Observation Period as the baseline and the total seizure frequency per 28 days of the Weeks, 12, 24, 32, 40, 52 and 52 LOCF as the post-treatment value. Percentage change in total seizure frequency was calculated as follows: [100 x (post-treatment value - baseline)/ baseline]. Seizures analyzed other than tonic-atonic seizures included: Partial seizure frequency, Absence seizure, Atypical absence seizure, Myoclonic seizure, Tonic seizure, Tonic-clonic seizure, Atonic seizure, and Unclassified epileptic seizure. This data was based on the diary data collected for 7 days after each visit. Seizure frequency was counted based on the classification established by the ILAE. The diary recorder monitored the participant and recorded the seizure diary in a consistent manner.
Time Frame: Baseline (Observation period in Study 304), Week 12, Week 24, Week 32, Week 40, Week 52 and Week 52 LOCF
Population: Efficacy Analysis Set included all participants with evaluable efficacy data.
Measure: Median (Full Range); unit: Percent Change in Seizure Frequency
Arm/Group | Rufinamide
Number analyzed (Participants) | 45
Percent Change in Seizure Frequency
  Partial Seizure Week 12: number analyzed (Participants) | 7
  Partial Seizure Week 12 | -95 [-100 to 255.6]
  Partial Seizure Week 24: number analyzed (Participants) | 5
  Partial Seizure Week 24 | -80.9 [-100 to 303.2]
  Partial Seizure Week 32: number analyzed (Participants) | 5
  Partial Seizure Week 32 | -70.5 [-100 to 30.2]
  Partial Seizure Week 40: number analyzed (Participants) | 5
  Partial Seizure Week 40 | -85.7 [-100 to -42.4]
  Partial Seizure Week 52: number analyzed (Participants) | 5
  Partial Seizure Week 52 | -77.3 [-100 to -61.8]
  Partial Seizure Week 52 LOCF: number analyzed (Participants) | 7
  Partial Seizure Week 52 LOCF | -77.3 [-100 to 189.2]
  Absence Seizure Week 12: number analyzed (Participants) | 1
  Absence Seizure Week 12 | -87.7 [-87.7 to -87.7]
  Absence Seizure Week 24: number analyzed (Participants) | 1
  Absence Seizure Week 24 | -100 [-100 to -100]
  Absence Seizure Week 32: number analyzed (Participants) | 1
  Absence Seizure Week 32 | -100 [-100 to -100]
  Absence Seizure Week 40: number analyzed (Participants) | 1
  Absence Seizure Week 40 | -100 [-100 to -100]
  Absence Seizure Week 52: number analyzed (Participants) | 1
  Absence Seizure Week 52 | -100 [-100 to -100]
  Absence Seizure Week 52 LOCF: number analyzed (Participants) | 1
  Absence Seizure Week 52 LOCF | -100 [-100 to -100]
  Atypical Absence Seizure Week 12: number analyzed (Participants) | 24
  Atypical Absence Seizure Week 12 | -86.7 [-100 to 54.7]
  Atypical Absence Seizure Week 24: number analyzed (Participants) | 22
  Atypical Absence Seizure Week 24 | -92.85 [-100 to 185.7]
  Atypical Absence Seizure Week 32: number analyzed (Participants) | 22
  Atypical Absence Seizure Week 32 | -92.3 [-100 to 209.2]
  Atypical Absence Seizure Week 40: number analyzed (Participants) | 21
  Atypical Absence Seizure Week 40 | -100 [-100 to 219.3]
  Atypical Absence Seizure Week 52: number analyzed (Participants) | 21
  Atypical Absence Seizure Week 52 | -100 [-100 to 737.2]
  Atypical Absence Seizure Week 52 LOCF: number analyzed (Participants) | 24
  Atypical Absence Seizure Week 52 LOCF | -100 [-100 to 737.2]
  Myoclonic Seizure Week 12: number analyzed (Participants) | 13
  Myoclonic Seizure Week 12 | -100 [-100 to 228.8]
  Myoclonic Seizure Week 24: number analyzed (Participants) | 13
  Myoclonic Seizure Week 24 | -100 [-100 to 64.4]
  Myoclonic Seizure Week 32: number analyzed (Participants) | 13
  Myoclonic Seizure Week 32 | -100 [-100 to 435.6]
  Myoclonic Seizure Week 40: number analyzed (Participants) | 13
  Myoclonic Seizure Week 40 | -100 [-100 to 117.6]
  Myoclonic Seizure Week 52: number analyzed (Participants) | 13
  Myoclonic Seizure Week 52 | -100 [-100 to 368.2]
  Myoclonic Seizure Week 52 LOCF: number analyzed (Participants) | 14
  Myoclonic Seizure Week 52 LOCF | -100 [-100 to 368.2]
  Tonic Seizure Week 12 | -35.4 [-100 to 175.2]
  Tonic Seizure Week 24: number analyzed (Participants) | 42
  Tonic Seizure Week 24 | -37.85 [-100 to 138.5]
  Tonic Seizure Week 32: number analyzed (Participants) | 41
  Tonic Seizure Week 32 | -49.4 [-100 to 83.5]
  Tonic Seizure Week 40: number analyzed (Participants) | 40
  Tonic Seizure Week 40 | -47.05 [-100 to 833.2]
  Tonic Seizure Week 52: number analyzed (Participants) | 39
  Tonic Seizure Week 52 | -36.4 [-100 to 110.2]
  Tonic Seizure Week 52 LOCF | -46.2 [-100 to 110.2]
  Tonic-clonic Seizure Week 12: number analyzed (Participants) | 8
  Tonic-clonic Seizure Week 12 | -61.55 [-100 to 300]
  Tonic-clonic Seizure Week 24: number analyzed (Participants) | 7
  Tonic-clonic Seizure Week 24 | -44.1 [-100 to 300]
  Tonic-clonic Seizure Week 32: number analyzed (Participants) | 7
  Tonic-clonic Seizure Week 32 | -22.6 [-100 to 700]
  Tonic-clonic Seizure Week 40: number analyzed (Participants) | 7
  Tonic-clonic Seizure Week 40 | -46.7 [-100 to 1100]
  Tonic-clonic Seizure Week 52: number analyzed (Participants) | 7
  Tonic-clonic Seizure Week 52 | -35.5 [-100 to 700]
  Tonic-clonic Seizure Week 52 LOCF: number analyzed (Participants) | 8
  Tonic-clonic Seizure Week 52 LOCF | -38.1 [-100 to 700]
  Atonic Seizure Week 12: number analyzed (Participants) | 16
  Atonic Seizure Week 12 | -60.35 [-100 to 29]
  Atonic Seizure Week 24: number analyzed (Participants) | 15
  Atonic Seizure Week 24 | -84.3 [-100 to 189.2]
  Atonic Seizure Week 32: number analyzed (Participants) | 14
  Atonic Seizure Week 32 | -100 [-100 to 20.5]
  Atonic Seizure Week 40: number analyzed (Participants) | 14
  Atonic Seizure Week 40 | -67.2 [-100 to 261.4]
  Atonic Seizure Week 52: number analyzed (Participants) | 14
  Atonic Seizure Week 52 | -67.55 [-100 to 526.5]
  Atonic Seizure Week 52 LOCF: number analyzed (Participants) | 16
  Atonic Seizure Week 52 LOCF | -67.55 [-100 to 526.5]
  Unclassified Seizure Week 12: number analyzed (Participants) | 1
  Unclassified Seizure Week 12 | -100 [-100 to -100]
  Unclassified Seizure Week 24: number analyzed (Participants) | 1
  Unclassified Seizure Week 24 | 6932.3 [6932.3 to 6932.3]
  Unclassified Seizure Week 32: number analyzed (Participants) | 1
  Unclassified Seizure Week 32 | -100 [-100 to -100]
  Unclassified Seizure Week 40: number analyzed (Participants) | 1
  Unclassified Seizure Week 40 | -100 [-100 to -100]
  Unclassified Seizure Week 52: number analyzed (Participants) | 1
  Unclassified Seizure Week 52 | -100 [-100 to -100]
  Unclassified Seizure Week 52 LOCF: number analyzed (Participants) | 1
  Unclassified Seizure Week 52 LOCF | -100 [-100 to -100]

5. Secondary Outcome: Percentage of Participants Who Achieved 100%, 75%, 50% or 25% Reduction in Tonic-Atonic Seizure Frequency (Responders)
Description: Categorized percent change in Tonic-atonic seizure frequency per 28 Days by visit relative to the baseline (Observation Phase in Study 304) was determined based on the diary data collected for 7 days after each visit. The Efficacy Analysis Set was used.
Time Frame: Week 12, Week 24, Week 32, Week 40, Week 52 and Week 52 LOCF
Population: Efficacy Analysis Set included all participants with evaluable efficacy data.
Measure: Number; unit: Percentage of participants
Arm/Group | Rufinamide
Number analyzed (Participants) | 46
Percentage of participants
  Week 12 100% Reduction - Yes | 6.5
  Week 12 100% Reduction - No | 93.5
  Week 12 75% Reduction - Yes | 17.4
  Week 12 75% Reduction - No | 82.6
  Week 12 50% Reduction - Yes | 43.5
  Week 12 50% Reduction - No | 56.5
  Week 12 25% Reduction - Yes | 71.7
  Week 12 25% Reduction - No | 28.3
  Week 24 100% Reduction - Yes | 2.3
  Week 24 100% Reduction - No | 97.7
  Week 24 75% Reduction - Yes | 11.6
  Week 24 75% Reduction - No | 88.4
  Week 24 50% Reduction - Yes | 39.5
  Week 24 50% Reduction -No | 60.5
  Week 24 25% Reduction - Yes | 65.1
  Week 24 25% Reduction - No | 34.9
  Week 32 100% Reduction - Yes | 2.4
  Week 32 100% Reduction - No | 97.6
  Week 32 75% Reduction - Yes | 19
  Week 32 75% Reduction - No | 81
  Week 32 50% Reduction - Yes | 47.6
  Week 32 50% Reduction - No | 52.4
  Week 32 25% Reduction - Yes | 66.7
  Week 32 25% Reduction - No | 33.3
  Week 40 100% Reduction - Yes | 4.9
  Week 40 100% Reduction - No | 95.1
  Week 40 75% Reduction - Yes | 17.1
  Week 40 75% Reduction - No | 82.9
  Week 40 50% Reduction - Yes | 48.8
  Week 40 50% Reduction - No | 51.2
  Week 40 25% Reduction - Yes | 61
  Week 40 25% Reduction - No | 39
  Week 52 100% Reduction - Yes | 5
  Week 52 100% Reduction - No | 95
  Week 52 75% Reduction - Yes | 20
  Week 52 75% Reduction -No | 80
  Week 52 50% Reduction - Yes | 37.5
  Week 52 50% Reduction - No | 62.5
  Week 52 25% Reduction - Yes | 60
  Week 52 25% Reduction - No | 40
  Week 52 (LOCF) 100% Reduction - Yes | 8.7
  Week 52 (LOCF) 100% Reduction - No | 91.3
  Week 52 (LOCF) 75% Reduction - Yes | 21.7
  Week 52 (LOCF) 75% Reduction -No | 78.3
  Week 52 (LOCF) 50% Reduction - Yes | 39.1
  Week 52 (LOCF) 50% Reduction - No | 60.9
  Week 52 (LOCF) 25% Reduction - Yes | 63
  Week 52 (LOCF) 25% Reduction - No | 37

6. Secondary Outcome: Percentage of Participants With An Increase In Tonic-Atonic Seizure Frequency
Description: Number of participants with an increase in Tonic-atonic seizure frequency per 28 Days by visit relative to the baseline (Observation Phase in Study 304) was determined based on the diary data collected for 7 days after each visit. The Efficacy Analysis Set was used.
Time Frame: Week 12, Week 24, Week 32, Week 40, Week 52 and Week 52 LOCF
Population: Efficacy Analysis Set included all participants with evaluable efficacy data.
Measure: Number; unit: Percentage of participants
Arm/Group | Rufinamide
Number analyzed (Participants) | 46
Percentage of participants
  Week 12 Increase - Yes | 21.7
  Week 12 Increase - No | 78.3
  Week 24 Increase - Yes | 23.3
  Week 24 Increase - No | 76.7
  Week 32 Increase - Yes | 16.7
  Week 32 Increase - No | 83.3
  Week 40 Increase - Yes | 9.8
  Week 40 Increase - No | 90.2
  Week 52 Increase - Yes | 22.5
  Week 52 Increase -No | 77.5
  Week 52 LOCF Increase - Yes | 19.6
  Week 52 LOCF Increase - No | 80.4

ADVERSE EVENTS:
Time Frame: From date of first dose up to 15 days after the last dose of study treatment, up to approximately 2 years and 10 months
Description: Safety analysis set included all treated participants.
Arm/Group | Rufinamide
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 9/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rufinamide (N=54)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Status epilepticus (Nervous system disorders) | 2 (4)
Dental caries (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rufinamide (N=54)
Contusion (Injury, poisoning and procedural complications) | 12 (22)
Skin laceration (Injury, poisoning and procedural complications) | 5 (9)
Eyelid injury (Injury, poisoning and procedural complications) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Mouth injury (Injury, poisoning and procedural complications) | 4 (4)
Platelet count decreased (Investigations) | 3 (3)
Weight decreased (Investigations) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Status epilepticus (Nervous system disorders) | 22 (158)
Somnolence (Nervous system disorders) | 14 (17)
Dizziness (Nervous system disorders) | 3 (4)
Conjunctivitis allergic (Eye disorders) | 3 (4)
Pyrexia (General disorders) | 5 (12)
Insomnia (Psychiatric disorders) | 6 (6)
Agitation (Psychiatric disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 13 (27)
Constipation (Gastrointestinal disorders) | 9 (10)
Dental caries (Gastrointestinal disorders) | 7 (8)
Stomatitis (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7)
Nasopharyngitis (Infections and infestations) | 26 (61)
Influenza (Infections and infestations) | 11 (15)
Upper respiratory tract infection (Infections and infestations) | 6 (16)
Bronchitis (Infections and infestations) | 5 (9)
Gastroenteritis (Infections and infestations) | 5 (5)
Pharyngitis (Infections and infestations) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other